CLINICAL TRIAL: NCT04898868
Title: Investigation on the Effects of Delayed Cord Clamping on Maternal and Neonatal Outcomes: Part I. Association Between Blood Volume, the Interval From Delivery to Cord Clamping, and Number of Umbilical Cord Milking
Brief Title: Association Between Blood Volume, the Interval From Delivery to Cord Clamping, and Number of Umbilical Cord Milking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tai-Ho Hung, Attending physician, Dept of Obs & Gyn, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201901045A3
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Pregnancy Related; Umbilical Cord Issue; Placental Transfusion
Keywords: Delayed umbilical cord clamping; umbilical cord milking
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Intervention Model Description: The investigators will recruit 80 women normal term pregnancy; 40 with vaginal delivery and 40 with elective CS for previous CS or fetal malpresentation.
  Participants will be randomized into 4 groups: group 1, vaginal delivery with cord blood spontaneous drainage; group 2, vaginal delivery with cord milking; group 3, CS with cord blood spontaneous drainage; group 4, CS with cord milking. In women allocated to groups of cord blood spontaneous drainage, two clamps will placed at 4 finger breadths from the infant's abdomen and cut between two clamps. The newborns will be taken care by the nurse after delivery. The clamp on the placenta site will be removed and record the drainage time and amount of cord blood to a measuring glass. In women allocated to groups of cord milking group, the umbilical cord will be squeezed several times, 5 seconds between each squeezing, to collect cord blood after delivery. The number of cord milking and the volume of blood collected will be recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vaginal delivery with cord blood spontaneous drainage (Experimental): In women allocated to groups of cord blood spontaneous drainage, two clamps will placed at 4 finger breadths from the infant's abdomen and cut between two clamps immediately after delivery of the baby. The clamp on the placental site will be removed and the drainage time and amount of cord blood to a measuring glass will be recorded.
  Interventions: Procedure: cord blood spontaneous drainage
- vaginal delivery with cord milking (Experimental): In women allocated to groups of cord milking group, two clamps will placed at 4 finger breadths from the newborn's abdomen and cut between two clamps immediately after delivery of the baby. The newborns will be taken care by the nurse. The clamp on the placental site will be removed, then the umbilical cord will be squeezed several times, 5 seconds between each squeezing, to collect cord blood in a measuring glass. The number of cord milking and the volume of blood collected will be recorded.
  Interventions: Procedure: Umbilical cord miking
- CS with cord blood spontaneous drainage (Experimental): In women allocated to groups of cord blood spontaneous drainage, two clamps will placed at 4 finger breadths from the infant's abdomen and cut between two clamps immediately after delivery of the baby. The clamp on the placental site will be removed and the drainage time and amount of cord blood to a measuring glass will be recorded.
  Interventions: Procedure: cord blood spontaneous drainage
- CS with cord milking (Experimental): In women allocated to groups of cord milking group, two clamps will placed at 4 finger breadths from the newborn's abdomen and cut between two clamps immediately after delivery of the baby. The newborns will be taken care by the nurse. The clamp on the placental site will be removed, then the umbilical cord will be squeezed several times, 5 seconds between each squeezing, to collect cord blood in a measuring glass. The number of cord milking and the volume of blood collected will be recorded.
  Interventions: Procedure: Umbilical cord miking

INTERVENTIONS:
Procedure: cord blood spontaneous drainage — In women allocated to groups of cord blood spontaneous drainage, two clamps will placed at 4 finger breadths from the infant's abdomen and cut between two clamps after delivery of the baby. The clamp on the placental site will be removed and the drainage time and amount of cord blood to a measuring glass will be recored.
  Arms: CS with cord blood spontaneous drainage; vaginal delivery with cord blood spontaneous drainage
Procedure: Umbilical cord miking — In women allocated to groups of cord milking group, two clamps will placed at 4 finger breadths from the newborn's abdomen and cut between two clamps immediately after delivery of the baby. The clamp on the placental site will be removed, then the umbilical cord will be squeezed several times, 5 seconds between each squeezing, to collect cord blood in a measuring glass. The number of cord milking and the volume of blood collected will be recorded.
  Arms: CS with cord milking; vaginal delivery with cord milking

SUMMARY:
Delayed umbilical cord clamping (DCC), usually 1-3 minutes, is reported to be beneficial for term and preterm infants. Nevertheless, there are reasons that urge us to reevaluate the effect of DCC. First, most prior studies were conducted on American and European women. The benefits of DCC in the infants born to Asian women is not clear. Second, neonates born to Asian mothers usually have lower birth weights and placental weights compared to the neonates and placentas of American and European women. The optimal duration of DCC in Asian women remains undetermined. The objective of this study is to determine the association between the blood volume collected and the interval from delivery to cord clamping and number of umbilical cord milking in women with normal term pregnancies with vaginal delivery or elective cesarean delivery (CS). Results form this study will help us determine the optimal duration of DCC or numbers of cord milking in our population in the following studies.

DETAILED DESCRIPTION:
Delayed umbilical cord clamping (DCC), usually 1-3 minutes, is reported to be beneficial for term and preterm infants. In term infants, DCC increases hemoglobin levels at birth and improves iron stores in the first several months of life, which may have a favorable effect on development outcomes. In preterm infants, the benefits of DCC include improved transitional circulation, better establishment of red blood cell volume, decreased need for blood transfusion, and lower incidence of necrotizing enterocolitis and intraventricular hemorrhage. DCC was not associated with increased risk of postpartum hemorrhage or increased blood loss at delivery, nor was it associated with the need for blood transfusion. Three is a small increase in the incidence of jaundice that requires phototherapy in infants undergoing DCC. Given the benefits of most newborns, a number of professional organizations recommends DCC in term and preterm infants, when feasible.

There are reasons that urge us to reevaluate the effect of DCC in our population. First, most prior studies were conducted on American and European women. The benefits of DCC in the infants born to Asian women is not clear. Second, neonates born to Asian mothers usually have lower birth weights and placental weights compared to the neonates and placentas of American and European women. The optimal duration of DCC in Asian women remains undetermined. With the aforementioned reasons, the investigators will conduct a study to clarify the effects of DCC and umbilical cord milking on maternal and neonatal outcomes in Taiwanese women. Our objective is to determine the association between the blood volume collected and the interval from delivery to cord clamping and number of umbilical cord milking in women with normal term pregnancies with vaginal delivery or elective cesarean delivery (CS);.

ELIGIBILITY:
Inclusion Criteria:

* Women with a normal singleton term pregnancy (37-41 weeks of gestation) and preparing for vaginal delivery
* Women with a normal singleton term pregnancy (37-41 weeks of gestation) and preparing for CS for previous CS or fetal malpresentation

Exclusion Criteria:

* Pregnancies complicated by gestational hypertensive disorders, diabetes mellitus, gestational diabetes mellitus, placenta previa, multiple gestation, fetal growth restriction, fetal anomalies (chromosomal or structural), and reassuring fetal heart rate tracing during delivery.
* Women plan to store her cord blood in a cord blood bank.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Blood volume | delivery of the baby
  Total cord blood volume collected with spontaneous drainage or cord milking

SECONDARY OUTCOMES:
Hemoglobin difference | Change from admission for delivery to the next day after delivery
  The difference of maternal hemoglobin level before and after delivery
Hematocrit difference | Change from admission for delivery to the next day after delivery
  The difference of maternal hematocrit level before and after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Ho Hung, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Taipei Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kugelman A, Borenstein-Levin L, Riskin A, Chistyakov I, Ohel G, Gonen R, Bader D. Immediate versus delayed umbilical cord clamping in premature neonates born < 35 weeks: a prospective, randomized, controlled study. Am J Perinatol. 2007 May;24(5):307-15. doi: 10.1055/s-2007-981434. Epub 2007 May 21. PMID 17516307
- [Background] Takami T, Suganami Y, Sunohara D, Kondo A, Mizukaki N, Fujioka T, Hoshika A, Akutagawa O, Isaka K. Umbilical cord milking stabilizes cerebral oxygenation and perfusion in infants born before 29 weeks of gestation. J Pediatr. 2012 Oct;161(4):742-7. doi: 10.1016/j.jpeds.2012.03.053. Epub 2012 May 12. PMID 22578578
- [Background] Rabe H, Reynolds G, Diaz-Rossello J. Early versus delayed umbilical cord clamping in preterm infants. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003248. doi: 10.1002/14651858.CD003248.pub2. PMID 15495045
- [Background] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Background] Fogarty M, Osborn DA, Askie L, Seidler AL, Hunter K, Lui K, Simes J, Tarnow-Mordi W. Delayed vs early umbilical cord clamping for preterm infants: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Jan;218(1):1-18. doi: 10.1016/j.ajog.2017.10.231. Epub 2017 Oct 30. PMID 29097178
- [Background] Tarnow-Mordi W, Morris J, Kirby A, Robledo K, Askie L, Brown R, Evans N, Finlayson S, Fogarty M, Gebski V, Ghadge A, Hague W, Isaacs D, Jeffery M, Keech A, Kluckow M, Popat H, Sebastian L, Aagaard K, Belfort M, Pammi M, Abdel-Latif M, Reynolds G, Ariff S, Sheikh L, Chen Y, Colditz P, Liley H, Pritchard M, de Luca D, de Waal K, Forder P, Duley L, El-Naggar W, Gill A, Newnham J, Simmer K, Groom K, Weston P, Gullam J, Patel H, Koh G, Lui K, Marlow N, Morris S, Sehgal A, Wallace E, Soll R, Young L, Sweet D, Walker S, Watkins A, Wright I, Osborn D, Simes J; Australian Placental Transfusion Study Collaborative Group. Delayed versus Immediate Cord Clamping in Preterm Infants. N Engl J Med. 2017 Dec 21;377(25):2445-2455. doi: 10.1056/NEJMoa1711281. Epub 2017 Oct 29. PMID 29081267
- [Background] Kaempf JW, Tomlinson MW, Kaempf AJ, Wu Y, Wang L, Tipping N, Grunkemeier G. Delayed umbilical cord clamping in premature neonates. Obstet Gynecol. 2012 Aug;120(2 Pt 1):325-30. doi: 10.1097/AOG.0b013e31825f269f. PMID 22825092
- [Background] Committee Opinion No. 684: Delayed Umbilical Cord Clamping After Birth. Obstet Gynecol. 2017 Jan;129(1):1. doi: 10.1097/AOG.0000000000001860. PMID 28002310
- [Background] Perry IJ, Beevers DG, Whincup PH, Bareford D. Predictors of ratio of placental weight to fetal weight in multiethnic community. BMJ. 1995 Feb 18;310(6977):436-9. doi: 10.1136/bmj.310.6977.436. PMID 7873949
- [Background] Jones J, Stevens CE, Rubinstein P, Robertazzi RR, Kerr A, Cabbad MF. Obstetric predictors of placental/umbilical cord blood volume for transplantation. Am J Obstet Gynecol. 2003 Feb;188(2):503-9. doi: 10.1067/mob.2003.19. PMID 12592263